CLINICAL TRIAL: NCT01348971
Title: Effects of Oral Nitrate During Coronary Artery Bypass Surgery
Brief Title: Coronary Artery Bypass and Nitrate Oral Supplementation
Acronym: CABANOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Eddie Weitzberg, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: KI-101
Record Dates: First submitted 2011-05-04; First posted 2011-05-06 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Coronary Artery Disease
Keywords: sodium nitrate; coronary artery bypass surgery; ischemia-reperfusion; myocardial injury
MeSH Terms: conditions — Coronary Artery Disease | interventions — sodium nitrate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium nitrate (Experimental): Preoperative oral administration of sodium nitrate. 700 mg the night before surgery and 700 mg three hours before surgery
  Interventions: Dietary Supplement: Sodium nitrate
- Placebo (Placebo Comparator): Preoperative oral administration of sodium chloride the night before surgery and three hours before surgery
  Interventions: Other: Sodium chloride

INTERVENTIONS:
Dietary Supplement: Sodium nitrate — Preoperative oral administration of sodium nitrate. 700 mg the night before surgery and 700 mg three hours before surgery
  Arms: Sodium nitrate
Other: Sodium chloride — Preoperative oral administration of sodium chloride the night before surgery and three hours before surgery
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether oral sodium nitrate administration prior to coronary artery bypass surgery can reduce perioperative levels of troponin T. In addition, plasma and urine surrogate markers of renal, hepatic and brain injury will be monitored.

DETAILED DESCRIPTION:
Nitric oxide (NO) is an important mediator in the cardiovascular system and has been shown to have protective properties in ischemia-reperfusion injury. Inorganic nitrate, an oxidation product from endogenous NO production and also a constituent in green leafy vegetables, can be recycled, via nitrite, back to bioactive NO in the body. Recent research has shown beneficial effects of nitrate and nitrite in animal models of myocardial ischemia-reperfusion injury. Moreover, dietary nitrate reduces blood pressure and oxygen cost during exercise in humans.

During coronary bypass surgery the heart undergoes ischemia-reperfusion injury and troponin T is most often released from the myocardium. The aim of the present study is to investigate if preoperative inorganic nitrate, in doses easily achievable from the diet, can affect troponin T release as well as other surrogate markers of injury to the liver, kidneys and the brain. In addition, plasma and urine samples will be collected for markers of oxidative stress and inflammation (sCRP and cytokines). Patients planned for bypass surgery who give their written informed consent will, the night before surgery, get a standardized, low-nitrate meal where after they receive sodium nitrate on two occasions preoperatively; the night before and in the morning before surgery. Plasma and urine samples will be collected at various time points up to 72 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coronary artery bypass surgery
* Over 18 years of age

Exclusion Criteria:

* Over 80 years of age
* Pregnancy
* Reoperation
* Intended heart valve or additional surgery
* Angina or troponin release above 45 nmol/L < 48 hours before surgery
* Medication with organic nitrates/nitrites < 24 hours before surgery
* Medication with glibenclamide or corticosteroids
* Significant renal, pulmonary or hepatic disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Troponin T release over the perioperative 72-hour period. | 72 hours

SECONDARY OUTCOMES:
Troponin T release over the perioperative 24-hour period. | 24 h
Creatinine kinase myocardial fraction (CKMB) release over the perioperative 72-hour period | 72 hours
Creatinine kinase myocardial fraction (CKMB) release over the perioperative 24-hour period | 24 hours
Pro Brain natriuretic peptide (proBNP) release over the perioperative 72-hour period. | 72 hours
Aspartate aminotransferase (AST) release over the perioperative 72-hour period. | 72 hours
Alaninaminotransferas (ALAT) release over the perioperative 72-hour period. | 72 hours
Alkaline phosphatase (ALP) release over the perioperative 72-hour period. | 72 hours
Bilirubin release over the perioperative 72-hour period | 72 hours
Creatinine release over the perioperative 72-hour period | 72 h
Cystatin C release over the perioperative 72-hour period | 72

CONTACTS AND LOCATIONS:
Overall Officials: Eddie T Weitzberg, MD,PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Eriksson KE, Eidhagen F, Liska J, Franco-Cereceda A, Lundberg JO, Weitzberg E. Effects of inorganic nitrate on ischaemia-reperfusion injury after coronary artery bypass surgery: a randomised controlled trial. Br J Anaesth. 2021 Oct;127(4):547-555. doi: 10.1016/j.bja.2021.06.046. Epub 2021 Aug 14. PMID 34399982